CLINICAL TRIAL: NCT03556514
Title: Follow-up for Locking Plate Fixaion of Distal Radius Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-05-009AC
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2017-06

CONDITIONS: Distal Radius Fracture
Keywords: Locking Plate Fixaion
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current status of the disease under study. Including natural history, disease prognosis.

Distal radial fractures (DRF, distal radius fractures) are the most common fractures, allowing the user to lock the steel plate to accelerate the recovery of the wrist, but related injuries such as the triangular fibrocartilage cartilage complex (TFCC) tear or distal radius ulna joint (DRUJ) ligament tear with DRUJ instability requires time fixed or further repair surgery. If these issues are ignored, there will be weakness in the future. The ulnar shortening commonly used by hand surgeons is to improve the damage of TFCC or DRUJ instability. In the case of distal radial fracture combined with DRUJ instability, it is not clear that the distal radial fracture combined with DRUJ instability patients has long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient following for at least one year

Exclusion Criteria:

* (1) Injury or arthritis before; (2) Open fractures, or more wounds require surgery

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute distal humerus fracture after interlocking plate fixation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-05-09 (Estimated); Study Completion 2019-05-09 (Estimated)

PRIMARY OUTCOMES:
4-Item Pain intensity Measure | 5 seconds
  Each item is scored 0-10(0=no pain;10=pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Pan Wang, M.D.,Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan